CLINICAL TRIAL: NCT06922357
Title: A Phase I/II, Open-label, Multi-centre Study Evaluating the Safety,Tolerability,Pharmacokinetic (PK), Pharmacodynamics, and Preliminary Efficacy of HRS-6719 in Patients With Advanced/Metastatic Solid Tumors With MTAP Deficiency
Brief Title: A Phase I/II of HRS-6719 in Patients With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6719-101
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-6719 (Experimental)
  Interventions: Drug: HRS-6719

INTERVENTIONS:
Drug: HRS-6719 — HRS-6719

SUMMARY:
This is a Phase I/II, multicenter, open-label clinical trial with dose escalation/dose expansion/efficacy expansion phases, designed to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic (PK/PD) profiles, and antitumor efficacy characteristics of HRS-6719 in patients with MTAP-deficient advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in the study and sign an informed consent form;
2. Aged 18-75 years, male or female eligible；
3. ECOG performance status score of 0-1；
4. Expected survival ≥12 weeks；
5. Patients with histologically or cytologically confirmed advanced malignant solid tumors who meet one of the following criteria:Disease progression or intolerance after receiving adequate standard therapy; Lack of standard treatment options;Currently ineligible for standard therapy；
6. Ability to provide sufficient fresh or archived tumor tissue specimens；
7. Adequate function of vital organs；
8. Effective contraception must be used during the trial. For women of childbearing potential, a negative pregnancy test within 7 days prior to the first dose is required。

Exclusion Criteria:

1. History of other malignant tumors within the past 5 years；
2. Received systemic anti-tumor therapy within 4 weeks prior to the first study dose.
3. Surgical procedures requiring tracheal intubation and general anesthesia were performed within 4 weeks before the first administration, diagnostic or surface surgery was performed within 1 week before the first administration, or elective surgery was expected during the trial.
4. The study received radical radiotherapy within 4 weeks before the first medication ; and received palliative radiotherapy within 2 weeks before the first medication.
5. Uncontrolled pleural, pericardial, or peritoneal effusions.
6. Severe cardiac diseases occurring within 6 months prior to the first dose.
7. Arterial/venous thrombosis within 6 months before the first dose.
8. Clinically significant bleeding symptoms or predisposition within 3 months prior to the first dose.
9. Active infection or fever of unknown origin > 38.5 ° C was present within 4 weeks before the first administration of the study
10. History of immunodeficiency.
11. Active hepatitis B or C.
12. Diseases affecting drug absorption/transport (e.g., malabsorption syndromes).
13. A history of severe allergic reactions to HRS-6719 and its main components was known or suspected, or there was a history of delayed allergic reactions, eczema or asthma that could not be controlled by topical corticosteroids.
14. Use of strong CYP3A4/P-gp inhibitors/inducers within 5 half-lives before the first dose.
15. Adverse events (AEs) from prior anti-tumor therapy not resolved to CTCAE v5.0 ≤ Grade 1.
16. Patients with interstitial pneumonia or interstitial lung disease, or previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or clinically significant pulmonary fibrosis, persistent pneumonia, pneumonia caused by drug or radiotherapy, congenital pneumonia, or chest CT scan found any evidence of active pneumonia.
17. Through medical history or CT examination, it was found that there was active pulmonary tuberculosis infection within 1 year before enrollment, or more than 1 year ago, there was a history of active pulmonary tuberculosis infection but no formal treatment.
18. Live attenuated vaccines administered within 4 weeks before the first dose or planned during the study.
19. Other factors potentially compromising study safety or data integrity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
Maximum tolerable dose (MTD) | 21 Days (first cycle)
Recommended dose for phase II (RP2D) | through phase I completion, an average of 1 years
Incidence and severity of AE | from Day1 to 30 days after last dose

SECONDARY OUTCOMES:
Relative bioavailability after meals on an empty stomach | through phase I completion, an average of 1 years
ORR | 12 months after the last subject was enrolled in the group
DOR | 12 months after the last subject was enrolled in the group
DCR | 12 months after the last subject was enrolled in the group
TTR | 12 months after the last subject was enrolled in the group
PFS | 12 months after the last subject was enrolled in the group
OS | 1 Year after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided